CLINICAL TRIAL: NCT06080399
Title: Could Psycho-bio-social Context and Personality be a Predictive Factor of Quality of Life Amelioration After Continuous Subcutaneous Apomorphine Infusion in Parkinson's Disease Patients? - PERSO-PERF Study
Brief Title: Personality and Quality of Life Amelioration After Continuous Subcutaneous Apomorphine Infusion in Parkinson's Disease
Acronym: PERSO-PERF
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: ELIVIE France (Unknown); EVER Pharma France SAS (Unknown); NHC SAS, France (Unknown); Orkyn' (Industry); ETPARK Association, Toulouse, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0401
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; personality dimensions; TCI; CSAI; second-line treatment; quality of life
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Continuous subcutaneous apomorphine infusion (CSAI) — the CSAI proposed in the usual healthcare pathway of each PD patients included

SUMMARY:
Since our previous study has shown that some personality dimensions were associated with Quality of Life (QoL) amelioration after Deep Brain Stimulation (DBS) in Parkinson's disease (PD), the investigators aim to evaluate the impact of personality dimensions on therapeutic response after another second-line treatment: the continuous subcutaneous apomorphine infusion (CSAI). Moreover, the investigators would like to evaluate the potential evolution of personality dimensions through CSAI. The investigators also aim to evaluate other bio-psycho-social factors (representations of the disease, ways of copying and social support) influence on QoL amelioration after DBS.

DETAILED DESCRIPTION:
As Parkinson's disease (PD) progresses, the onset of motor and non-motor fluctuations alters patients Quality of Life (QoL). Second-line treatments can then be proposed: either the implantation of deep brain electrodes (Deep Brain Stimulation of the Sub-Thalamic Nuclei (DBS-STN)), or the drug approach (continuous subcutaneous infusion of apomorphine or continuous intrajejunal infusion of levodopa/carbidopa).

To date, no randomized double-blind trial has compared the efficacy and adverse effects of these different types of second-line treatments. There is therefore no clearly defined predictive factor that could predict better efficacy of these second-line treatments in patients, or the occurrence of adverse effects leading to discontinuation of these treatments.

The choice of treatment must consider patients specific personal needs as well as their clinical phenotype, this constitutes the major challenge of personalized medicine. Thus, personality, which reflects the way a person thinks, reflects, acts and behaves in different situations, appears to be a possible predictive criterion for QoL improvement after second-line treatments.

Indeed, using the Temperament and Character Inventory (TCI) self-questionnaire, the investigators have shown that two personality dimensions of the TCI ("Novelty Seeking" and "Cooperativeness") appeared to be predictive of QoL amelioration in PD patients after DBS-STN. Thus, the use of this personality questionnaire, the TCI, enables better prediction of patients therapeutic response after DBS-STN. It could also be useful to predict therapeutic response after other second-line treatments such as continuous subcutaneous infusion of apomorphine. In this study, the investigators therefore propose to evaluate the impact of personality dimensions on therapeutic response after the introduction of this infusion therapy.

Investigators carried out a preliminary exploratory study (PSYCHO-PERF study - ClinicalTrials.gov NCT03793491) which showed a significant association between a personality dimension of the TCI ("Reward Dependence") and QoL improvement after six months of continuous subcutaneous infusion of apomorphine in 33 PD patients (article in preparation). This suggests that patients with high Reward Dependence scores may be good candidates for continuous subcutaneous infusion of apomorphine. However, these results need to be confirmed on a larger scale, by means of a multicenter study.

Hence, some TCI personality dimensions in PD patients could be predictive of QoL improvement after second-line treatment. Thus, before proposing a second-line treatment, in the context of personalized medicine, personality assessment could be one of the criteria to choose between these different treatments.

However, the investigators are aware that PD patients personality can only partly explain the therapeutic response. For this reason, the investigators also wish to include in our study other psycho-bio-social factors (social representations of the disease and treatments, coping strategies and social support perceived by patients) that may influence QoL improvement following treatment.

In a more exploratory context, the investigators would also like to assess changes in TCI personality dimensions of PD patients following treatment with continuous subcutaneous infusion of apomorphine, since changes in mood and/or behavior have already been observed. If a change is observed, the investigators will determine whether this change is associated with clinical and demographic data prior to the continuous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patients as defined by the United Kingdom Parkinson's disease Brain Bank (UKPDSBB) criteria and aged from 40 to 75 years old (included)
* Patients with motor fluctuations and/or invalidating dyskinesia and awaiting CSAI establishment in the context of their usual care for PD
* Patients affiliated to a social security system

Exclusion Criteria:

* Patients presenting an atypical parkinsonian syndrome Patients having a Deep Brain Stimulation
* Patients with a psychiatric disease such as bipolar disorder or delusions linked to a dopaminergic psychosis
* Patients presenting a cognitive deficit attested by a score to the Montreal Cognitive Assessment inferior to 24, solely during the inclusion (baseline - V0)
* Patient with a serious pathology (e.g. cancer) or a health condition which could interfere with the assessment of their quality of life, at the discretion of the investigator upon inclusion
* Patients under guardianship, curatorship or safeguard of justice
* Patients under exclusion period from another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: parkinson's disease patients receiving CSAI
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the link between personality dimensions in baseline and QoL amelioration after six months | 6 months
  to evaluate the link between personality dimensions in baseline and QoL amelioration after six months of CSAI in PD patients, the coefficients of linear regressions between the scores of the different TCI personality dimensions at V0 (explicative variables) and the percentage of global QoL amelioration (Total PDQ-39 scores) (response variable) at V6 will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: CHRISTINE BREFEL COURBON, Principal Investigator — University Hospital, Toulouse
Locations (10):
- France (10):
  - Chu de Lyon, Bron
  - Hopital Gabriel Montpied, Clermont-Ferrand
  - Chu de Grenoble, Grenoble
  - Chu Limoges, Limoges
  - Chu de Nancy, Nancy
  - Chu de Nice, Nice
  - Chu de Poitiers, Poitiers
  - Chu de Rennes, Rennes
  - Chu de Rouen, Rouen
  - Chu de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Boussac M, Harroch E, Barthelemy C, Ory-Magne F, Leung C, Fabbri M, Arbus C, Brefel-Courbon C. Personality and quality-of-life improvement after apomorphine infusion in Parkinson's disease. Brain Commun. 2024 May 24;6(3):fcae181. doi: 10.1093/braincomms/fcae181. eCollection 2024. PMID 38846534